CLINICAL TRIAL: NCT03840330
Title: Effects of High-intensity Interval Circuit Training (HIICT) on the Cardiovascular and Functional Parameters of Aged Women
Brief Title: High-intensity Training for Improving Physical Performance of Aged Women
Acronym: AHIITATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, María Carrasco Poyatos, Principal Investigator, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HIICT-OW/16
Record Dates: First submitted 2018-09-05; First posted 2019-02-15 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Aging; Healthy; Cardiovascular Risk Factor; Physical Activity
Keywords: High-intensity interval training; Circuit training; Elderly; Functional capacity; VO2 max; Cardiovascular parameters
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: HIT; MIT; GC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-intensity interval training group (Experimental): Frequency: 2 days/weeks; Intensity: 16-18 Börg/85-100%VO2max; Recovery: Active; Duration: 1 hour.
  Interventions: Other: Experimental: High-intensity interval training group
- Moderate-intensity interval training group (Experimental): Frequency: 2 days/weeks; Intensity: 12-14 Börg/60-70% VO2max; Recovery: Active; Duration: 1 hour.
  Interventions: Other: Experimental: Moderate-intensity interval training group
- Control group (No Intervention): Maintain their normal daily activities throughout the sixteen-week experimental period.

INTERVENTIONS:
Other: Experimental: High-intensity interval training group — 16 weeks of High-intensity interval training
  Arms: High-intensity interval training group
Other: Experimental: Moderate-intensity interval training group — 16 weeks of Moderate-intensity interval training
  Arms: Moderate-intensity interval training group

SUMMARY:
This study evaluates the adaptations on the functional capacity and cardiovascular in elderly after a physical activity program circuit training. The participants were divided into three groups: Circuit training based on high-intensity interval training group (HIICT), Circuit training at moderate intensity group (MICT) and Control group (CG).

DETAILED DESCRIPTION:
Three groups of participants (circuit training based on high-intensity interval training, circuit training at moderate intensity and not training group) will enter the study. The intervention will consist of a physical exercise program in day centers.

Intensity progression will be encouraged according to the rate of perceived exertion. Progression of exertion will be "very hard", "extremely hard" and "maximal exertion" for HIT group, and "light", "somewhat hard" and "hard" for group. Assessment will be undertaken at two-time points: baseline and after 16 weeks of exercise training.

Assessment will include VO2 peak, functional capacity, health-related quality of life, cognitive state and daily physical activity.

ELIGIBILITY:
Inclusion Criteria:

1. Having 50 - 90 years old.
2. Not suffering chronic heart, respiratory or joint disease, taking medication or having a deteriorated level of mental health that could interfere in carrying out exercise programs.
3. Having 0 or 1 responses positive in the Physical Activity Readiness Questionnaire (ParQ). Only item 6, related to mild vascular diseases.
4. Being physically independent according to the scales Lawton and Brody, and Katz.

Exclusion Criteria:

1. Having uncontrolled arterial hypertension.
2. Having practiced during the previous 3 months or practicing at present a similar exercise to the one proposed in the study.
3. Attending sessions less than 80%.

Ages: 50 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 54 (Actual)
Dates: Start 2015-12-20 (Actual); Primary Completion 2016-02-01 (Actual); Study Completion 2016-06-20 (Actual)

PRIMARY OUTCOMES:
Analyses changes in maximum oxygen consumption (VO2max). | Pre and post after sixteen weeks of intervention
  A modified Balke treadmill protocol will be used to estimate aerobic capacity (VO2max).
Analyses changes in maximum oxygen consumption (VO2max). | Pre and post after sixteen weeks of intervention
  VO2max was assessed using the 6-Minute Walk Test. The participant should walk the longest distance possible in 6 minutes by walking continuously the 42 metres indicated on the floor. It measures the distance in meters

SECONDARY OUTCOMES:
Analyses changes in heart rate reached in ergometry. | Pre and post after sixteen weeks of intervention
  Analyses during modified Balke treadmill protocol
Analyses changes in blood pressure reached in ergometry. | Pre and post after sixteen weeks of intervention
  Analyses during modified Balke treadmill protocol
Analyses changes in maximum speed reached in ergometry. | Pre and post after sixteen weeks of intervention
  Analyses during modified Balke treadmill protocol
Analyses changes in duration test reached in ergometry. | Pre and post after sixteen weeks of intervention
  Analyses during modified Balke treadmill protocol
Analyses changes in fat percentage. | Pre and post after sixteen weeks of intervention.
  Fat percentage (%) was assessed using bioimpedance analysis (OMROM BF-306).
Analyses changes in body mass index (BMI). | Pre and post after sixteen weeks of intervention.
  BMI was assessed using bioimpedance analysis (OMROM BF-306).
Analyses changes in gait. | Pre and post after sixteen weeks of intervention.
  Gait was assessed using the Timed Up and Go Test. To stand up from a standard arms chair, walk 3 meters, turn back the cone walk back and sit down to the chair. The time in seconds is record.
Analyses changes in balance. | Pre and post after sixteen weeks of intervention.
  Balance was assessed using the One Leg Standing Test. This test consist in maintain one leg stance for as long as possible. The test was considered normal if the one leg standing time reached 30 seconds.
Analyses changes in lower body strength. | Pre and post after sixteen weeks of intervention.
  Lower body strength was assessed using the Sit To Stand 30. For the Sit To Stand 30, the participant consist in measures how many repetition the participant can to stand up and sit down during 30 seconds.
Analyses changes in upper body strength. | Pre and post after sixteen weeks of intervention.
  Upper body strength was assessed using the Arm Curl Test (30). For this test, the participant consist in measures how many repetition the participant can to curl up and curl down during 30 seconds.
Analyses changes in maximal handgrip strength. | Pre and post after sixteen weeks of intervention.
  To measure the amount of strength developed by each hand in kg.

OTHER OUTCOMES:
Analyses change in Self Assessed Physical Activity. | Pre and post after sixteen weeks of intervention.
  Physical activity was assessed using the Physical Activity Scale of the Elderly (PASE) questionnaire. The PASE is designed to assess physical activity in older persons. The total PASE score was computed by multiplying the amount of time spent in each activity (hours/week) or participation (yes/no) in an activity by empirically derived item weights and summing over all activities. PASE scores for this study ranged from 0 to 756 with higher scores indicating more physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Ismael Ballesta García, PhD. Student, Principal Investigator — Universidad de Almeria; María Carrasco Poyatos, PhD., Principal Investigator — Universidad de Almeria

REFERENCES:
- [Result] Wisloff U, Stoylen A, Loennechen JP, Bruvold M, Rognmo O, Haram PM, Tjonna AE, Helgerud J, Slordahl SA, Lee SJ, Videm V, Bye A, Smith GL, Najjar SM, Ellingsen O, Skjaerpe T. Superior cardiovascular effect of aerobic interval training versus moderate continuous training in heart failure patients: a randomized study. Circulation. 2007 Jun 19;115(24):3086-94. doi: 10.1161/CIRCULATIONAHA.106.675041. Epub 2007 Jun 4. PMID 17548726
- [Result] Guiraud T, Juneau M, Nigam A, Gayda M, Meyer P, Mekary S, Paillard F, Bosquet L. Optimization of high intensity interval exercise in coronary heart disease. Eur J Appl Physiol. 2010 Mar;108(4):733-40. doi: 10.1007/s00421-009-1287-z. PMID 19915859
- [Result] Huang SC, Wong MK, Lin PJ, Tsai FC, Fu TC, Wen MS, Kuo CT, Wang JS. Modified high-intensity interval training increases peak cardiac power output in patients with heart failure. Eur J Appl Physiol. 2014 Sep;114(9):1853-62. doi: 10.1007/s00421-014-2913-y. Epub 2014 Jun 1. PMID 24880226
- [Result] Ballesta Garcia I, Rubio Arias JA, Ramos Campo DJ, Martinez Gonzalez-Moro I, Carrasco Poyatos M. High-intensity Interval Training Dosage for Heart Failure and Coronary Artery Disease Cardiac Rehabilitation. A Systematic Review and Meta-analysis. Rev Esp Cardiol (Engl Ed). 2019 Mar;72(3):233-243. doi: 10.1016/j.rec.2018.02.015. Epub 2018 Apr 9. English, Spanish. PMID 29650445
- See also: Carrasco, M., Navarro, M.D., Martínez, I., Reche-Orenes, D. (2016). Daily physical activity impact in old women bone density and grip strength. Nutrición Hospitalaria, 33(6), 1305-1311. — http://scielo.isciii.es/scielo.php?script=sci_abstract&pid=S0212-16112016000600008
- See also: Carrasco, M., Martínez, I., Navarro, M.D. (2015). Daily physical activity and bone mineral density in older women. Revista Brasileira de Medicina do Esporte, 21(1), 22-26. — http://www.scielo.br/scielo.php?script=sci_arttext&pid=S1517-86922015000100022

DOCUMENTS (1):
  • Informed Consent Form (2010-02-10): https://cdn.clinicaltrials.gov/large-docs/30/NCT03840330/ICF_000.pdf